CLINICAL TRIAL: NCT04053114
Title: MOLecular Characterization and Treatment of THYroid Carcinoma on Struma Ovarii
Acronym: MOLTHYSO
Status: Withdrawn | Type: Observational
Why Stopped: Principal investigator left the investigational center and nobody took over.
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB2018-MOLTHYSO; MR 0016040319 (Other: Institut National des Données de Santé (INDS))
Record Dates: First submitted 2019-07-04; First posted 2019-08-12 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer
Keywords: Ovarian teratoma; struma ovarii; thyroid carcinoma; next generation sequencing
MeSH Terms: conditions — Ovarian Neoplasms; Teratoma, Ovarian; Struma Ovarii; Thyroid Neoplasms | interventions — DNA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Frozen or FFPE tumoral specimens suitable for DNA and RNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Retrospective cohort: Tissue samples
  Interventions: Other: DNA and RNA extraction from FFPE or frozen tissue sample

INTERVENTIONS:
Other: DNA and RNA extraction from FFPE or frozen tissue sample — Next generation sequencing (NGS)

SUMMARY:
Thyroid carcinoma on struma ovarii (TCSO) is a rare ovarian tumor, derivate from monodermic teratomas. It represents about 0.01% of overall ovarian tumours, and 5 to 10% of struma ovarii. The diagnosis is histologic and retrospective after pelvic surgery. Because of its rarity, the treatment of TCSO is not consensual and should be validated in multidisciplinary team involved in rare ovarian carcinoma. TCSO should be taken care of as a thyroid carcinoma, in case of relapse, with systemic treatment, as tyrosine kinase inhibitor (TKI), without any clinical trial proving this benefit. Indeed, molecular profiles and genomic expression is unknown, because of studies with few patients (less than 10) contrary to thyroid carcinomas with the TCGA genomic classification. The study purposes are the outcome of the patients after the first treatment and the comparison of the genomic profil in next generation sequencing (NGS) with TCGA thyroid carcinoma profile. Thus, the treatment could be tailored, confirming the same therapy as in thyroid carcinoma.

DETAILED DESCRIPTION:
This is a retrospective cohort with collection of tissues samples (FFPE or frozen), including female patients >18-year-old treated in French between 2009 and 2016 for a thyroid carcinoma on struma ovarii. Clinical data and tissues will be centralized for assessment. One of the endpoint is the description of the population (such as baseline clinical and pathologist characteristics, first treatment, survival, treatment relapse) ; the other endpoint is the comparison between the genomic profile of the tumor tissues obtained in NGS and those of the thyroid carcinomas obtained from the TCGA.

ELIGIBILITY:
Inclusion Criteria:

* Alive patients,
* Age > 18 years,
* Treatment in France for a TCSO, proven by an histologic diagnosis and registered in the " rare malignant gynecologic tumors " network.

Exclusion Criteria:

- Patient lost to follow up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French women older than 18 years old with a TCSO registered in the French " Rare malignant gynecologic tumors " network from 2007 to 2017.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Treatment description | Between first treatment and last follow up, assessed up to 100 months
  Description of the previous treatment for the TCSO (first treatment and relapse) in the retrospective cohort

CONTACTS AND LOCATIONS:
Overall Officials: Anne FLOQUET, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No